CLINICAL TRIAL: NCT05756387
Title: Improving Chronic Nocturnal Noninvasive Ventilation: a Multimodality Approach
Acronym: NOCTIVENT
Status: Recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: University of Twente (Other); Löwenstein BV (Unknown); Vivisol (Other); Sencure BV (Unknown)
Responsible Party: Sponsor
Other Study IDs: 16013
Record Dates: First submitted 2023-02-13; First posted 2023-03-06 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Chronic Respiratory Failure; Non-invasive Ventilation
Keywords: Monitoring
MeSH Terms: interventions — Noninvasive Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- COPD patients with Chronic Respiratory Failure
  Interventions: Device: Non-invasive ventilation

INTERVENTIONS:
Device: Non-invasive ventilation — NIV as in standard care

SUMMARY:
The aim of the data collection is to create an advanced reliable method to remotely monitor patient on chronic home non-invasive ventilation (NIV), both regarding ventilatory efficacy and patient comfort, both in the hospital and at home by assessing gas exchange, lung mechanics and the interaction between the patient and the ventilator.

For this purpose, we will set-up of databank of synchronously acquired datasets of already standard care monitored parameters during NIV (transcutaneous monitoring of gas exchange; ventilator data including data on PVA), and newly non-invasively acquired data on patient effort (EMG, patient ratings) and lung (hyper)inflation (EIT), during the set-up and follow-up of standard care chronic NIV.

DETAILED DESCRIPTION:
Can be provided on request as the registry rules are no in Dutch

ELIGIBILITY:
Inclusion Criteria:

* COPD patients indicated for chronic home NIV

Exclusion Criteria:

* not able to read the written information and/or sign the informed consent form
* no possibility to perfrom measurements at home

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: COPD patients with chronic hypercapnic respiratory failure needing chronic NIV will be included
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Gas exchange | baseline
  Transcutaneous monitoring of gas exchange
Gas exchange | 2 months
  Transcutaneous monitoring of gas exchange
Gas exchange | 4 months
  Transcutaneous monitoring of gas exchange
Gas exchange | 6 months
  Transcutaneous monitoring of gas exchange
Patient comfort | baseline
  Patient comfort assessed by VAS scale
Patient comfort | 2 months
  Patient comfort assessed by VAS scale
Patient comfort | 4 months
  Patient comfort assessed by VAS scale
Patient comfort | 6 months
  Patient comfort assessed by VAS scale
AECOPD | 2 months, 4 months, 6 months
  Acute exacerbations of COPD (defines as deterioration of symptoms requiring a course of/increase in Prednisolone dose and/or antibiotics)
AECOPD | 2 months
  Acute exacerbations of COPD (defines as deterioration of symptoms requiring a course of/increase in Prednisolone dose and/or antibiotics)
AECOPD | 4 months
  Acute exacerbations of COPD (defines as deterioration of symptoms requiring a course of/increase in Prednisolone dose and/or antibiotics)
Hospitalisations for AECOPD | 6 months
  Hospitalisations for acute exacerbations of COPD
Sleep quality | 2 months
  Sleep quality assessing sleep depth and sleep stages
Sleep quality | 4 months
  Sleep quality assessing sleep depth and sleep stages
Sleep quality | 6 months
  Sleep quality assessing sleep depth and sleep stages

CONTACTS AND LOCATIONS:
Overall Officials: Marieke L Duiverman, Principal Investigator — University Medical Center Groningen
Locations (1):
- UMCG, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided